CLINICAL TRIAL: NCT02616263
Title: Muscle, Joint and Movement Deterioration Contributing to Neuropathic Forefoot Deformity
Brief Title: Metatarsal Phalangeal Joint Deformity Progression - R01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Mary Hastings, PT, DPT, ATC, Professor of Physical Therapy, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: DK107809
Record Dates: First submitted 2015-11-18; First posted 2015-11-26 (Estimated); Results first posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus (DM)
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Foot Intervention (Experimental): The intervention is a progressive, home based exercise program aimed to increase ankle and foot plantarflexion muscle strength, increase ankle dorsiflexion and toe flexion range of motion, and to retrain individuals to dorsiflex the ankle while keeping the toes in a neutral position. A trained physical therapist with experience working with older adults with diabetes and foot specific complications will monitor and progress the exercise program assuring participant safety and maximizing exercise benefit.
  Interventions: Other: Foot exercise
- Shoulder Intervention (Active Comparator): Participants will be trained in a progressive home exercise program that includes passive stretching of end range shoulder flexion and external rotation and a tailored dose of active shoulder motion.
  Interventions: Other: Shoulder exercise

INTERVENTIONS:
Other: Foot exercise
  Arms: Foot Intervention
Other: Shoulder exercise
  Arms: Shoulder Intervention

SUMMARY:
The purpose of this research study is to determine the relationships between foot muscle, foot motion, and toe deformity. Results from this investigation will help the investigators to understand what contributes to foot deformities and the role of the foot muscles in the development of foot deformities. This could potentially guide treatment options focusing on strengthening the foot muscles to prevent or reduce the risk of developing a foot deformity.

DETAILED DESCRIPTION:
The long term goal of this research is to reduce the incidence of lower extremity amputation in people with diabetes mellitus and peripheral neuropathy. It is hypothesized that muscle, joint, and movement deterioration associated with diabetes and peripheral neuropathy contribute to metatarsophalangeal joint (MTPJ) hyperextension deformity. MTPJ deformity results in excessive plantar stress on the insensitive forefoot, leading to ulceration and amputation. However, the specific cause of MTPJ deformity is not clear. The overall goal of this proposal is to identify the causes of MTPJ deformity and examine the ability of a targeted foot specific intervention to de-couple diabetes related mechanisms from MTPJ deformity and progression, following participants for 3 years. The investigators hypothesize that the cause of MTPJ deformity is an interaction of the accumulation of advanced glycation end products, muscle deterioration, limited joint mobility and compensatory movement strategies.

The specific aims are to determine:

1. relationships between advanced glycation end products, intrinsic foot muscle volume, limited ankle dorsiflexion joint mobility, MTPJ hyperextension movement pattern, and MTPJ alignment;
2. estimate the effect of a foot specific intervention on the MTPJ extension alignment and
3. determine progression of MTPJ deformity and the predictors of progression over three years.

The following will be collected on participants with diabetes mellitus and peripheral neuropathy and monitored over three years to understand the causes and progression of MTPJ deformity:

1. Skin intrinsic florescence to measure advanced glycation end product accumulation which increases collagen cross-linking and is associated with peripheral neuropathy, limited joint mobility, and muscle deterioration.
2. Magnetic resonance images to measure intrinsic foot muscle deterioration that precedes extrinsic foot muscle deterioration as a result of distal to proximal peripheral neuropathy. The muscle imbalance of weak intrinsic foot muscles, the only muscles able to flex the MTPJ, in the presence of relatively stronger extrinsic toe extensors, results in a force couple that hyperextends the MTPJ.
3. Kinematic and computed tomography measurement of foot and ankle joint positions to examine mobility and movement patterns that contribute to repeated and extreme MTPJ hyperextension during daily activities.

The investigators believe advanced glycation end products lead to limited ankle joint dorsiflexion. As a result, there is increased reliance on the extensor digitorum longus to assist in dorsiflexing the stiff ankle joint during activities like sit to stand. This study will have profound implications for reducing risk for skin breakdown and amputation by helping to understand and treat the causes of acquired neuropathic foot deformities. A successful foot specific intervention that improves MTPJ alignment will provide a non-invasive option to halt or slow the cascade of events leading to major lower extremity amputation, while improving function and minimizing disability.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus (DM)
* Diabetic peripheral neuropathy

Exclusion Criteria:

* active plantar ulcers, unable to ambulate or complete required testing, anyone who have amputations of their lower extremity (>1 toe), weigh more than 400 lbs, pregnant, have metal implants or pace makers (incompatible with MRI), greater than 75 years old, Subjects with other causes of PN (lumbar radiculopathy, microvascular disease, alcoholic/HIV/chemotaxic neuropathy), on dialysis, with peripheral arterial disease (ABI<0.9 or >1.3), with fixed MTPJ deformity (excursion <30 degrees active/passive), acute shoulder pain or disability that would prevent participation in shoulder specific intervention (i.e. severe shoulder pain >6/10, rotator cuff tear, upper extremity surgery, thoracic outlet syndrome);

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03; Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary K Hastings, PT,DPT,MSCI, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Other researchers may contact us to get access to the data but we will not be placing the data in a repository

REFERENCES:
- [Background] Harris-Hayes M, Schootman M, Schootman JC, Hastings MK. The Role of Physical Therapists in Fighting the Type 2 Diabetes Epidemic. J Orthop Sports Phys Ther. 2020 Jan;50(1):5-16. doi: 10.2519/jospt.2020.9154. Epub 2019 Nov 28. PMID 31775555
- [Background] Hastings MK, Commean PK, Chen L, Zellers JA, Sinacore DR, Baker JC. Qualitative study of musculoskeletal tissues and their radiographic correlates in diabetic neuropathic foot deformity. Foot (Edinb). 2021 Jun;47:101777. doi: 10.1016/j.foot.2021.101777. Epub 2021 May 3. PMID 33957525
- [Background] Holmes CJ, Hastings MK. The Application of Exercise Training for Diabetic Peripheral Neuropathy. J Clin Med. 2021 Oct 28;10(21):5042. doi: 10.3390/jcm10215042. PMID 34768562
- [Background] Zellers JA, Commean PK, Chen L, Mueller MJ, Hastings MK. A limited number of slices yields comparable results to all slices in foot intrinsic muscle deterioration ratio on computed tomography and magnetic resonance imaging. J Biomech. 2021 Dec 2;129:110750. doi: 10.1016/j.jbiomech.2021.110750. Epub 2021 Sep 13. PMID 34555631
- [Background] Zellers JA, Eekhoff JD, Walk RE, Hastings MK, Tang SY, Lake SP. Human Achilles tendon mechanical behavior is more strongly related to collagen disorganization than advanced glycation end-products content. Sci Rep. 2021 Dec 17;11(1):24147. doi: 10.1038/s41598-021-03574-4. PMID 34921194
- [Result] Zellers JA, Mueller MJ, Commean PK, Chen L, Jeong HJ, Hastings MK. Multi-System Factors Associated with Metatarsophalangeal Joint Deformity in Individuals with Type 2 Diabetes. J Clin Med. 2020 Apr 3;9(4):1012. doi: 10.3390/jcm9041012. PMID 32260124
- [Result] Hastings MK, Jeong HJ, Sorensen CJ, Zellers JA, Chen L, Bohnert KL, Snozek D, Mueller MJ. Relationships within and between lower and upper extremity dysfunction in people with diabetes. Foot (Edinb). 2020 Sep;44:101680. doi: 10.1016/j.foot.2020.101680. Epub 2020 Mar 30. PMID 32679515
- [Result] Jeong HJ, Mueller MJ, Zellers JA, Hastings MK. Midfoot and ankle motion during heel rise and gait are related in people with diabetes and peripheral neuropathy. Gait Posture. 2021 Feb;84:38-44. doi: 10.1016/j.gaitpost.2020.11.013. Epub 2020 Nov 16. PMID 33264731
- [Result] Jeong HJ, Mueller MJ, Zellers JA, Yan Y, Hastings MK. Heel Rise and Non-Weight-Bearing Ankle Plantar Flexion Tasks to Assess Foot and Ankle Function in People With Diabetes Mellitus and Peripheral Neuropathy. Phys Ther. 2021 Jul 1;101(7):pzab096. doi: 10.1093/ptj/pzab096. PMID 33735386
- [Result] Zellers JA, Bernhardson HJ, Jeong HJ, Commean PK, Chen L, Mueller MJ, Hastings MK. Association of toe-extension movement pattern magnitude and variability during three functional tasks with diabetic foot complications. Clin Biomech (Bristol). 2021 May;85:105371. doi: 10.1016/j.clinbiomech.2021.105371. Epub 2021 May 3. PMID 33965738
- [Result] Jeong HJ, Mueller MJ, Zellers JA, Commean PK, Chen L, Hastings MK. Body mass index and maximum available midfoot motion are associated with midfoot angle at peak heel rise in people with type 2 diabetes mellitus and peripheral neuropathy. Foot (Edinb). 2022 May;51:101912. doi: 10.1016/j.foot.2022.101912. Epub 2022 Feb 11. PMID 35255403
- [Result] Jeong HJ, Cha B, Zellers JA, Chen L, Hastings MK. Midfoot and ankle movement coordination during heel rise is disrupted in people with diabetes and peripheral neuropathy. Clin Biomech (Bristol). 2022 Jun;96:105662. doi: 10.1016/j.clinbiomech.2022.105662. Epub 2022 May 7. PMID 35569256
- [Result] Bohnert KL, Zellers JA, Jeong HJ, Chen L, York A, Hastings MK. Remote Research: Resources, Intervention Needs, and Methods in People with Diabetes and Peripheral Neuropathy. J Diabetes Sci Technol. 2023 Jan;17(1):52-58. doi: 10.1177/19322968221103610. Epub 2022 Jun 30. PMID 35770988
- [Derived] Youmans NJ, Vaidya RS, Chen L, Jeong HJ, York A, Commean PK, Hastings MK, Zellers JA. Rate of tarsal and metatarsal bone mineral density change in adults with diabetes mellitus and peripheral neuropathy: a longitudinal study. J Foot Ankle Res. 2023 Feb 13;16(1):6. doi: 10.1186/s13047-023-00606-2. PMID 36782282

RESULTS

PARTICIPANT FLOW:
Groups:
- Foot Intervention: The intervention is a progressive, home based exercise program aimed to increase ankle and foot plantarflexion muscle strength, increase ankle dorsiflexion and toe flexion range of motion, and to retrain individuals to dorsiflex the ankle while keeping the toes in a neutral position. A trained physical therapist with experience working with older adults with diabetes and foot specific complications will monitor and progress the exercise program assuring participant safety and maximizing exercise benefit.
  Foot exercise
- Shoulder Intervention: Participants will be trained in a progressive home exercise program that includes passive stretching of end range shoulder flexion and external rotation and a tailored dose of active shoulder motion.
  Shoulder exercise
Period: Baseline to 6 Month (Intervention Phase)
Arm/Group | Foot Intervention | Shoulder Intervention
Started | 29 | 31
Completed | 28 | 28
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Lost to Follow-up | 1 | 0
Period: 6 Month to 1.5 Year
Arm/Group | Foot Intervention | Shoulder Intervention
Started | 28 | 28
Completed | 26 | 25
Not Completed | 2 | 3
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1
Period: 1.5 Year to 3+ Year Follow up
Arm/Group | Foot Intervention | Shoulder Intervention
Started | 26 | 25
Completed | 22 | 23
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Foot Intervention | Shoulder Intervention | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 12 | 21
  >=65 years | 20 | 19 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.48 (8.05) | 66.55 (4.14) | 67 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 34
  Male | 14 | 12 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 10 | 16
  White | 21 | 21 | 42
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 26 | 27 | 53
  Unknown or not reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 29 | 31 | 60
Foot Joint Deformity [Mean (Standard Deviation); unit: Degrees]
  2nd Metatarsophalangeal Joint Hyperextension | 54.7 (12.3) | 51.4 (13.3) | 53.0 (12.8)
  Calcaneal Pitch | 21.5 (6.6) | 18.5 (5.3) | 20.0 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Metatarsal Phalangeal Joint Angle (Degrees) in People With Diabetes From Baseline and at a 3-year Period
Description: The angle between the 2nd metatarsal and the proximal phalanx will be measured at baseline and again at the 3-years
Time Frame: Three years
Population: 23 participants in each group completed 3 year follow up testing (average follow up time was 3.6 yrs due to COVID pause in human research testing) to assess the effect of the foot intervention on metatarsophalangeal joint extension alignment.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Foot Intervention | Shoulder Intervention
Number analyzed (Participants) | 23 | 23
degrees | 0.8 (9.3) | -0.1 (8.2)

ADVERSE EVENTS:
Time Frame: Through study completion, on average 3.6 years
Description: Adverse event were collected systematically through standardized questions answered during 3 month follow up phone calls or during study visits (e.g. falls, skin breakdown, foot pain, shoulder pain, changes in medical conditions, or new medical conditions). Unexpected adverse events were recorded when information was volunteered or discovered (e.g. failure to answer follow up phone calls resulted in a search of the social security web site to identify of participants were deceased).
Arm/Group | Foot Intervention | Shoulder Intervention
All-Cause Mortality (participants affected / at risk) | 1/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 12/29 | 19/31
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Foot Intervention (N=29) | Shoulder Intervention (N=31)
Falls (General disorders) | 5 (6) | 6 (7) — Participant report of falls during follow up phone calls or visits
Pain (General disorders) | 0 (0) | 4 (4) — Report of foot or shoulder pain
Foot skin breakdown (Skin and subcutaneous tissue disorders) | 7 (12) | 9 (17) — any cut, abrasion, sore on the foot

LIMITATIONS AND CAVEATS:
We excluded individuals with more severe foot deformity limiting generalizability of the study findings.

There were some delays in final time point assessment and participant attrition due to Covid-19 related restrictions on human subjects research around the final time point

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT02616263/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-02): https://cdn.clinicaltrials.gov/large-docs/63/NCT02616263/ICF_001.pdf